CLINICAL TRIAL: NCT02876055
Title: Prospective, Randomized Controlled Trial Comparing Analgesic Efficacy of Single Injection vs. Continuous Interscalene Blockade vs. Local Infiltration Analgesia for Patients Undergoing Primary Total Shoulder Arthroplasty
Brief Title: Analgesic Efficacy of Interscalene Nerve Block Versus Local Infiltration Analgesia Following Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jason K. Panchamia, D.O., Instructor in Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-009646
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Pain, Postoperative
Keywords: Nerve Block/methods; Pain, Postoperative/prevention & control; Anesthetics, Local/administration & dosage; Brachial Plexus/ultrasonography; Shoulder Pain/prevention & control
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single shot interscalene nerve block (Active Comparator): An interscalene nerve block will be performed under continuous live ultrasound guidance, obtaining visualization of the roots or trunks of the brachial plexus in between the anterior and middle scalene muscles. 15 to 20 mL of Bupivacaine 0.5% with 1:200,000 Epinephrine will be administered.
  Interventions: Drug: Single shot interscalene nerve block
- Continuous interscalene nerve block (Active Comparator): An interscalene nerve block and delivery of a catheter will be performed under continuous live ultrasound guidance, obtaining visualization of the roots or trunks of the brachial plexus in between the anterior and middle scalene muscles.
  Initial loading bolus includes 15 to 20 mL of Bupivacaine 0.5% with 1:200,000 Epinephrine. After surgery, the continuous interscalene nerve block catheter will be loaded in the post-anesthesia care unit (PACU) with bupivacaine 0.2% 10 milliliters (mL), and then an infusion will be initiated of bupivacaine 0.2% at 8 to 10 mL per hour.
  Interventions: Drug: Continuous interscalene nerve block
- Local Infiltration Analgesia (LIA) (Experimental): The LIA group will utilize weight based dosing of Ropivacaine as part of a "cocktail" solution containing ropivacaine, epinephrine, ketorolac, and normal saline 0.9%. Patients will receive a total volume of 120 mL injected strategically in the periarticular structures by the surgeon. This is a one-time injection. This will occur after implantation of the final prostheses, but prior to closure of the fascia.
  Interventions: Drug: Local Infiltration Analgesia (LIA)

INTERVENTIONS:
Drug: Single shot interscalene nerve block — Peripheral regional anesthesia nerve block - Single shot interscalene nerve block
  Other Names: Interscalene brachial plexus block
  Arms: Single shot interscalene nerve block
Drug: Continuous interscalene nerve block — Peripheral regional anesthesia nerve block - continuous catheter interscalene nerve block
  Other Names: Interscalene brachial plexus block
  Arms: Continuous interscalene nerve block
Drug: Local Infiltration Analgesia (LIA) — Injection of local anesthetic into the peri-articular tissues and intra-articular capsule in a systematic approach for orthopedic surgery
  Other Names: Arthroplasty Block; Peri-articular Injection
  Arms: Local Infiltration Analgesia (LIA)

SUMMARY:
Total shoulder arthroplasty (TSA) is considered to be a major surgical procedure resulting in severe postoperative pain, especially in the first 48 hours after surgery. The use of interscalene brachial plexus nerve block remains the cornerstone for analgesia following shoulder surgery; however, with the advent of local infiltration analgesia (LIA), there has been increasing interest in its use for total joint arthroplasty.

Since the benefits of local infiltration analgesia within a comprehensive multi-modal analgesia clinical pathway have yet to be established for total shoulder arthroplasty, the Investigators plan to assess and compare analgesia outcomes between three intervention groups: single shot interscalene brachial plexus block (SISB), continuous interscalene brachial plexus block (CISB), and local infiltration analgesia (LIA).

ELIGIBILITY:
Inclusion criteria:

1. Adult patients with an American Society of Anesthesiologists (ASA) physiological status I-III
2. Patients presenting for unilateral primary total shoulder arthroplasty (includes anatomic and reverse total shoulder arthroplasty).
3. Patients 18 years of age and older
4. Able to provide informed consent for him or herself

Exclusion Criteria:

1. Chronic pain syndromes such as fibromyalgia or complex regional pain syndrome
2. Chronic opioid use (>1 mos) with oral morphine equivalents (OME) >5 mg/day OR acute opioid use (< 1 mos) with OME > 30 mg/day.
3. Body mass index (BMI) > 45 kg/m2
4. Severe drug allergy* to medications used in this study, including non-steroidal anti-inflammatory drugs (i.e. celecoxib and ketorolac), and local anesthetics.
5. History of Malignant Hyperthermia.
6. Major systemic medical problems such as:

   * Pre-existing severe renal disorder defined as glomerular filtration rate (GFR) <50 units/m2 (if labs are available), currently on dialysis, or highly suspected based on history.
   * Severe hepatic disorder defined as current or past diagnosis of acute/subacute necrosis of liver, acute hepatic failure, chronic liver disease, cirrhosis (primary biliary cirrhosis), chronic hepatitis/toxic hepatitis, liver abscess, hepatic coma, hepatorenal syndrome, other disorders of liver
   * Pre-existing medical history of moderate to severe pulmonary disease (obstructive and/or restrictive), use of home oxygen, preoperative baseline oxygen saturation < 94% on room air, forced expiratory volume in 1 second (FEV 1) < 60% of predicted value (obstructive disease), vital capacity (VC) or total lung capacity (TLC) < 70% predicted value (restrictive disease).37
   * History of contralateral hemidiaphragmatic dysfunction (e.g., paralysis) or phrenic nerve injury.
7. Contraindication to a regional anesthesia technique (e.g., preexisting neuropathy+ in the operative extremity, coagulopathy, sepsis, infection at site of injection, uncooperative, refusal, anticoagulation medications not held within appropriate time frame per American Society of Regional Anesthesia (ASRA) guidelines.
8. Previous contralateral total shoulder replacement managed with regional anesthetic nerve block or periarticular injection/intraarticular injection within the previous 12 months.
9. Known to be currently pregnant or actively breastfeeding++

   • ++ Patients that have a previous history of menopause, hysterectomy, or tubal ligation will not be required to perform a pregnancy test.
10. Impaired cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Panchamia, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Interscalene Nerve Block: An interscalene nerve block and delivery of a catheter will be performed under continuous live ultrasound guidance, obtaining visualization of the roots or trunks of the brachial plexus in between the anterior and middle scalene muscles.
  Initial loading bolus includes 15 to 20 mL of Bupivacaine 0.5% with 1:200,000 Epinephrine. After surgery, the continuous interscalene nerve block catheter will be loaded in the post-anesthesia care unit (PACU) with bupivacaine 0.2% 10 milliliters (mL), and then an infusion will be initiated of bupivacaine 0.2% at 8 to 10 mL per hour.
  Continuous interscalene nerve block: Peripheral regional anesthesia nerve block - continuous catheter interscalene nerve block
Period: Overall Study
Arm/Group | Single Shot Interscalene Nerve Block | Continuous Interscalene Nerve Block | Local Infiltration Analgesia (LIA)
Started | 42 | 41 | 42
Completed | 42 | 41 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Continuous Interscalene Nerve Block: An interscalene nerve block and delivery of a catheter will be performed under continuous live ultrasound guidance, obtaining visualization of the roots or trunks of the brachial plexus in between the anterior and middle scalene muscles.
  Initial loading bolus includes 15 to 20 mL of Bupivacaine 0.5% with 1:200,000 Epinephrine. After surgery, the continuous interscalene nerve block catheter will be loaded in the PACU with bupivacaine 0.2% 10 milliliters (mL), and then an infusion will be initiated of bupivacaine 0.2% at 8 to 10 mL per hour.
  Continuous interscalene nerve block: Peripheral regional anesthesia nerve block - continuous catheter interscalene nerve block
- Total: Total of all reporting groups
Arm/Group | Single Shot Interscalene Nerve Block | Continuous Interscalene Nerve Block | Local Infiltration Analgesia (LIA) | Total
Number analyzed (Participants) | 42 | 41 | 42 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (13.1) | 68.1 (10.1) | 69.5 (8.9) | 68.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 17 | 61
  Male | 20 | 19 | 25 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 42 | 125
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (5.2) | 30.2 (5.7) | 30.9 (5.0) | 30.4 (5.3)
American Society of Anesthesiologists (ASA) Status [Count of Participants; unit: Participants] — ASA classification defines ASA I as a normal healthy patient, ASA II as a patient with a mild systemic disease without substantive functional limitations and an ASA III as a patient with a severe systemic disease with substantive functional limitations. A lower classification (I/II) is a more positive reflection of overall health compared to a higher classification (III).
  Participants
    ASA I/II | 28 | 26 | 27 | 81
    ASA III | 14 | 15 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Comparing Pain Intensity and Opioid-Related Adverse Effects Using Overall Benefit of Analgesia Score (OBAS).
Description: The OBAS score was calculated using the sum of the scores from six questions. OBAS ranges from 0 (best) to 28 (worst), where a low score indicates a high benefit to the subjects.
Time Frame: Post-Operative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single Shot Interscalene Nerve Block | Continuous Interscalene Nerve Block | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 42 | 41 | 42
score on a scale | 2 [1 to 4] | 0 [0 to 2] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Single Shot Interscalene Nerve Block vs Local Infiltration Analgesia (LIA); Test type: Superiority; p = 0.542, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Continuous Interscalene Nerve Block vs Local Infiltration Analgesia (LIA); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Single Shot Interscalene Nerve Block vs Continuous Interscalene Nerve Block; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to 3 months following last administration of study treatment for each subject.
Arm/Group | Single Shot Interscalene Nerve Block | Continuous Interscalene Nerve Block | Local Infiltration Analgesia (LIA)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 1/42
Other Adverse Events (participants affected / at risk) | 1/42 | 3/41 | 1/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Interscalene Nerve Block (N=42) | Continuous Interscalene Nerve Block (N=41) | Local Infiltration Analgesia (LIA) (N=42)
ICU admission (General disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Shot Interscalene Nerve Block (N=42) | Continuous Interscalene Nerve Block (N=41) | Local Infiltration Analgesia (LIA) (N=42)
Neurapraxia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02876055/Prot_SAP_000.pdf